CLINICAL TRIAL: NCT02624427
Title: Comparison of Intraocular Pressure Measured by Goldmann Applanation Tonometry and Dynamic Contour Tonometry vs. Corvis ST Tonometer
Brief Title: Goldmann Applanation Tonometry, Dynamic Contour Tonometry, and Corvis ST Tonometer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Corvis and DCT vs. GAT
Record Dates: First submitted 2015-11-27; First posted 2015-12-08 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Glaucoma
Keywords: Glaucoma; Intraocular Pressure
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glaucoma Eyes (Experimental): Measurement of intraocular pressure (IOP)
  Interventions: Device: Measurement of intraocular pressure (IOP)
- Healthy Eyes (Active Comparator): age-matched healthy eyes as controls will undergo Measurement of intraocular pressure (IOP)
  Interventions: Device: Measurement of intraocular pressure (IOP)

INTERVENTIONS:
Device: Measurement of intraocular pressure (IOP) — Measurement of IOP with the following devices: (1) Goldmann tonometer, (2) Dynamic Contour tonometer, and (3) Corvis ST tonometer

SUMMARY:
The study is investigating Intra ocular pressure (IOP) by Goldmann Applanation Tonometry, Dynamic Contour Tonometry, and the Corvis ST tonometer.

DETAILED DESCRIPTION:
The aim of the study is to approach the "true" Intra ocular pressure (IOP) by correlating the difference between IOP by Goldmann Applanation Tonometry to the IOP by Dynamic Contour Tonometry to the biomechanical parameters of the cornea measured by Corvis ST. Therefore the investigators gain new findings about the influence of the biomechanical corneal parameters on the IOP. In order to do so the investigators want to examine 50 Glaucoma eyes and 50 non-Glaucoma Eyes with Goldmann Applanation Tonometry, Dynamic Contour Tonometry, and Corvis ST.

ELIGIBILITY:
Inclusion Criteria for the glaucoma group:

* diagnosis of glaucoma
* 18 years old or older with no upper limit

Exclusion Criteria for the glaucoma group:

* IOP lowering surgery within the last 3 weeks
* any corneal surgery in the past
* bad fixation
* insufficient measurement quality with any of the study devices

Inclusion Criteria for the healthy control group:

* no diagnosis of glaucoma
* 18 years old or older with no upper limit

Exclusion Criteria for the healthy control group:

* any diagnosis of glaucoma
* IOP lowering surgery within the last 3 weeks
* any corneal surgery in the past
* bad fixation
* insufficient measurement quality with any of the study devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2015-12; Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Delta IOP | baseline
  IOP difference of Goldmann tonometer and Dynamic Contour tonometer

SECONDARY OUTCOMES:
Correlation of IOP difference of Goldmann tonometer and Dynamic Contour tonometer with biomechanical corneal properties measured by Corvis ST tonometer | baseline
  Corvis ST has an integrated high-speed Scheimpflug camera which records images on which basis the biomechanical corneal parameter are analyzed (corneal thickness in micrometers, corneal applications in millimeters, peak distance in millimeters, radius in millimeters, and deformation amplitude in millimeters). Those biomechanical parameters of the cornea will be correlated to the difference of the IOP measured by GAT and by DCT (GAT - DCT).

CONTACTS AND LOCATIONS:
Overall Officials: Jens Funk, MD PhD, Principal Investigator — UniversityHospital of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Center — http://www.usz.ch